CLINICAL TRIAL: NCT04494230
Title: Motor Proficiency in School Age ADHD: Contribution of Different Comorbidities
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Nilay Şahan, Hacettepe University, Hacettepe University
Other Study IDs: GO 18/694
Record Dates: First submitted 2020-07-28; First posted 2020-07-31 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2018-10

CONDITIONS: Attention Deficit Hyperactivity Disorder; Comorbidities and Coexisting Conditions; Motor Skills Disorders
Keywords: Attention Deficit Hyperactivity Disorder; comorbidity; motor skills
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Motor Skills Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Attention deficit hyperactivity disorder (ADHD) only: the diagnosis of ADHD
  Interventions: Behavioral: Motor Proficiency in School Age ADHD: Contribution of Different Comorbidities
- Attention deficit hyperactivity disorder (ADHD) andSpecificand: the diagnosis of ADHD and SLD
  Interventions: Behavioral: Motor Proficiency in School Age ADHD: Contribution of Different Comorbidities
- ADHD and oppositional defiant disorder (ODD): the diagnosis of ADHD and ODD
  Interventions: Behavioral: Motor Proficiency in School Age ADHD: Contribution of Different Comorbidities
- ADHD and Anxiety Disorder: the diagnosis of ADHD and Ank. Dis.
  Interventions: Behavioral: Motor Proficiency in School Age ADHD: Contribution of Different Comorbidities
- Typical Development Children: no mental symptoms described by their teachers or parents and showing healthy development
  Interventions: Behavioral: Motor Proficiency in School Age ADHD: Contribution of Different Comorbidities

INTERVENTIONS:
Behavioral: Motor Proficiency in School Age ADHD: Contribution of Different Comorbidities — to investigate whether motor skills, manual dexterity and visual perception differ in the presence of ADHD and comorbid psychiatric conditions in school-age boys by comparing them typical development children.

SUMMARY:
In this study, aged 6-10 years, male, right hand dominant, diagnosed with ADHD, accepting to take part in the study and applying to the Child and Adolescent Psychiatry Department between October 1, 2018 - October 1, 2019 were included in the research group.As for the control group, boys between 6-10 years of age with no mental symptoms described by their teachers or parents and showing healthy development were selected by convenience sampling method and snow ball method. Height and weight measurements of all the children participated in the study were performed. The sociodemographic data form prepared by the researchers was completed by both the research and the control group families.

In the sample, the Corners' Parent Scale- Revised Short Form (CPS-R:SF) was used to evaluate the severity of ADHD symptoms.The hand preferences of all participants in the research and control groups were evaluated with Edinburgh Handedness Inventory.Motor skills were evaluated with the 2nd Version of Bruininsky-Oseretsky Motor Competence Test (BOT-2).Hand skills were evaluated with the 9-Hole Peg Test.Visual perception skills were evaluated with 3rd Version of Visual Perception Test without Motor Ability (MVPT-3). Pediatric Quality of Life Inventory Parent Form were filled by the parents of children in the research and control groups for quality of life. In the study, there are five groups: ADHD, ADHD + Specific learning disorders, ADHD + Oppositional defiant disorder, ADHD + Anxiety Disorder and children with typical development group.

DETAILED DESCRIPTION:
In this study, aged 6-10 years, male, right hand dominant, diagnosed with ADHD, accepting to take part in the study and applying to the Child and Adolescent Psychiatry Department between October 1, 2018 - October 1, 2019 were included in the research group. A total of 106 children with head trauma or known neurological disease, clinically diagnosed as comorbid tic disorder, obsessive-compulsive disorder, psychotic disorder, mood disorder, conduct disorder, mental retardation, or autism spectrum disorder, or children previously excluded from physical therapy program were evaluated according to the research method. As for the control group; 30 boys between 6-10 years of age with no mental symptoms described by their teachers or parents and showing healthy development were selected by convenience sampling method and snow ball methodHeight and weight measurements of all the children participated in the study were performed. The sociodemographic data form prepared by the researchers was completed by both the research and the control group families.

In the sample, the Corners' Parent Scale- Revised Short Form (CPS-R:SF) was used to evaluate the severity of ADHD symptoms (Conners, 1997).

The hand preferences of all participants in the research and control groups were evaluated with Edinburgh Handedness Inventory.

Motor skills were evaluated with the 2nd Version of Bruininsky-Oseretsky Motor Competence Test (BOT-2). It is a standard test commonly used by physiotherapists to detect coarse and fine motor problems in children aged 4-21 years. It has both short and long form. The short form was used in our study. The short form of BOT-2 consists of 8 subtests: fine motor precision, fine motor integration, manual dexterity, bilateral coordination, balance, speed of movement and agility, upper extremity coordination and strength. Not only can the score of each subtest of the test be calculated separately but it can also be calculated as fine motor skill, gross motor skill, both fine and gross motor skill and total motor skill score.

Hand skills were evaluated with the 9-Hole Peg Test. The nine-hole Peg Test is a quick, simple and manual skill test that is particularly sensitive to changes in upper extremity performance. The test material consists of nine small rods made of standard sizes and nine perforated boards into which they are placed. In our study, insertion and removal periods for both dominant and nondominant hands were recorded separately.

Visual perception skills were evaluated with 3rd Version of Visual Perception Test without Motor Ability (MVPT-3). MVPT-3 is a fast, reliable test that tests visual perception without motor skills in children and adults (ages 4-65). The test consists of 65 questions and the first 40 questions were developed to test school-age children in terms of visual perception without motor skills as follows: visual discrimination (1-8), form constancy (9-13), visual memory-I (14-21), visual closure (22-34), visual differentiation (35-40). Total visual perception score and scores from each category were calculated separately. Pediatric Quality of Life Inventory Parent Form were filled by the parents of children in the research and control groups for quality of life. The scale has separate parent and child forms for the groups of 5-7 years, 8-12 years and 13-18 years. Scoring of the scale is done in 3 areas. Firstly, scale total score (STS) is calculated, and secondly, physical health total score (PHTS) is calculated. Thirdly, psychosocial health total score (PHTS) is calculated, which consists of calculating item scores evaluating emotional, social and school functionality. In the study, there are five groups: ADHD, ADHD + Specific learning disorders, ADHD + Oppositional defiant disorder, ADHD + Anxiety Disorder and children with typical development group.

ELIGIBILITY:
Inclusion Criteria:

* children aged 6-10 years, male, right hand dominant, diagnosed with ADHD, accepting to take part in the study and applying to the Child and Adolescent Psychiatry Department

Exclusion Criteria:

* with head trauma or known neurological disease, clinically diagnosed as comorbid tic disorder, obsessive-compulsive disorder, psychotic disorder, mood disorder, conduct disorder, mental retardation, or autism spectrum disorder, or children previously excluded from physical therapy program

Ages: 6 Years to 10 Years | Sex: Male
Age Groups: Child
Gender Based: Yes — school-aged male children
Study Population: children aged 6-10 years, male, right hand dominant
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
severity ADHD symptoms | 10 minutes
  the Corners' Parent Scale- Revised Short Form (CPS-R:SF) was used to evaluate the severity of ADHD symptoms. The scale whose Turkish adaptation study was made by Kaner et al. (2006) consists of 27 items. In CPS-R:SF, questions are answered on a 4-point Likert scale and high scores indicate the intensity of symptoms.
motor profiency | 40-45 minutes
  Motor skills were evaluated with the 2nd Version of Bruininsky-Oseretsky Motor Competence Test (BOT-2) (Bruininks, 1978). It is a standard test commonly used by physiotherapists to detect coarse and fine motor problems in children aged 4-21 years. It has both short and long form. The short form was used in our study. The short form of BOT-2 consists of 8 subtests: fine motor precision, fine motor integration, manual dexterity, bilateral coordination, balance, speed of movement and agility, upper extremity coordination and strength. Not only can the score of each subtest of the test be calculated separately but it can also be calculated as fine motor skill, gross motor skill, both fine and gross motor skill and total motor skill score.
hand skills | 10 minutes
  Hand skills were evaluated with the 9-Hole Peg Test. This questionnaire questions a hand or both hands used in daily life activities such as writing, drawing, ball throwing, using scissors, using a toothbrush, using a fork-free knife, using a spoon, sweeping with a broom handle, burning matches and opening boxes
visual perception | 30 minutes
  Visual perception skills were evaluated with 3rd Version of Visual Perception Test without Motor Ability (MVPT-3). MVPT-3 is a fast, reliable test that tests visual perception without motor skills in children and adults (ages 4-65). The test consists of 65 questions and the first 40 questions were developed to test school-age children in terms of visual perception without motor skills as follows: visual discrimination (1-8), form constancy (9-13), visual memory-I (14-21), visual closure (22-34), visual differentiation (35-40). Total visual perception score and scores from each category were calculated separately
quality of life | 15-20 minutes
  Quality of life were evaluated with Pediatric Quality of Life Inventory (PedsQL) aims to measure the overall quality of life in the 2-18 age group. The scale has separate parent and child forms for the groups of 5-7 years, 8-12 years and 13-18 years. Scoring of the scale is done in 3 areas. Firstly, scale total score (STS) is calculated, and secondly, physical health total score (PHTS) is calculated. Thirdly, psychosocial health total score (PHTS) is calculated, which consists of calculating item scores evaluating emotional, social and school functionality. The higher the total score of the scale is, the better the quality of life related to health is perceived

CONTACTS AND LOCATIONS:
Overall Officials: Nilay Şahan, PhD,PT, Principal Investigator — unaffilliated
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Goulardins JB, Marques JC, De Oliveira JA. Attention Deficit Hyperactivity Disorder and Motor Impairment. Percept Mot Skills. 2017 Apr;124(2):425-440. doi: 10.1177/0031512517690607. Epub 2017 Jan 31. PMID 28361657